CLINICAL TRIAL: NCT04269850
Title: Pilot Study of Fecal Microbiota Transplantation in Combination With Ruxolitinib and Steroids for Severe Acute Intestinal Graft-versus-host-disease After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Fecal Microbiota Transplantation With Ruxolitinib and Steroids as an Upfront Treatment of Severe Acute Intestinal GVHD
Acronym: JAK-FMT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Deputy Director for research, Raisa Gorbacheva Memorial Research Institute for Pediatric Oncology, Hematology and Transplantation Affiliation: St. Petersburg State Pavlov Medical University, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: tfm-gvhd-2019
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Intestinal GVHD
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT+ruxolitinib+steroids (Experimental): ruxolitinib 10 mg bid, fecal microbiota transplantation 2 caps/kg single dose, methylprednisone 0.5 mg/kg bid
  Interventions: Biological: allogeneic fecal microbiota; Drug: Ruxolitinib; Drug: Methylprednisone

INTERVENTIONS:
Biological: allogeneic fecal microbiota — Single dose of capsules with fecal transplant (capsules for adults - 400-815mg, for adolescents - 280-500mg, for children - 160-320mg) - 2 capsules/kg body weight, divided in two consecutive days Additional supportive therapy after FMT include omeprazole 40mg po, inulin 1gr x 4 times a day po, metoclopramide 40mg po.
Drug: Ruxolitinib — Ruxolitinib starting dose 10 mg bid. In case of grade 4 hematological toxicity dose can be reduced by 25-75%.
Drug: Methylprednisone — Methylprednisone starting dose 0.5 mg/kg bid IV or oral, with subsequent tapper by 0.1 mg/kg every 5 days.

SUMMARY:
Therapy of severe intestinal graft-versus-host disease (GVHD) despite the introduction of novel target agents is associated with worse outcome compared to the other forms. Response to steroids is observed only in about 10% of patients. The most promising approaches are JAK inhibition and fecal microbiota transplantation. In this pilot study we evaluate this combination treatment in the first line.

DETAILED DESCRIPTION:
Acute intestinal GVHD grade III-IV after allogeneic stem cell transplantation the form with low effectiveness of corticosteroids. Despite high response rate to systemic immunosupressive agents, long term survival in this group is poor due to recurrent septic episodes and gut colonization with multidrug resistant bacteria. Fecal microbiota transplantation (FMT) from a healthy allogeneic donor, allows to restore numerous local and systemic microbiota functions, including immunomodulation and thus to reduce/stop the manifestations of GVHD. The therapeutic mechanism of action of FMT is based on competition for nutrients between obligate and pathologic bacterial strains, direct growth inhibition of the pathological pathogens, host immune system modulation, especially T-reg homeostasis, through interaction with the normal microbiota.In this pilot trial we combine FMT with ruxolitinib and steroids, one of the most effective option for refractory GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-70 years
* Histologically confirmed gastrointestinal acute GVHD
* Grade III-IV gastrointestinal GVHD based on 2016 MAGIC criteria
* Ability for oral drug intake
* Signed informed consent

Exclusion Criteria:

* Requirement for oxigen and/or vasopressor support
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits,creatinine clearance < 60 mL/min
* Ongoing fluconazole therapy
* Any malignancy requiring systemic therapy at the time of enrollment
* Mixed chimerism at last evaluation
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Severe concurrent illness that can interfere with study procedures
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Overall survival | 365 days
  Time from treatment initiation to death or end of follow up

SECONDARY OUTCOMES:
Overal response rate | 100 days
  Evaluated with 2009 consensus criteria and 2016 severity grading on days +7,+28, +56, +100
Incidence of Adverse Events based on CTC AE 5.0 | 100 days
  Based on CTC AE 5.0
Infectious complications | 100 days
  Cumulative incidence of bacterial, viral and fungal infections
Time to steroid discontinuation | 100 days
  Time from treatment initiation to steroid cessation without GVHD flare
Time to ruxolitinib discontinuation | 365 days
  Time from treatment initiation to ruxolitinib cessation without GVHD flare
Time to systemic immunosuppression discontinuation | 365 days
  Time from treatment initiation to cessation of all systemic immunosupression without GVHD flare

CONTACTS AND LOCATIONS:
Overall Officials: Boris Afanasyev, Professor, Principal Investigator — Pavlov First Saint Petersburg State Medical University
Locations (1):
- Pavlov First Saint-Petersburg State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No